CLINICAL TRIAL: NCT06128291
Title: The Impact of Concomitant Posterior Colporrhaphy on Bowel Functions in Women Who Received Pelvic Organ Prolapse Repair
Brief Title: Concomitant Posterior Colporrhaphy on Bowel Functions in Pelvic Organ Prolapse Repair
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202303052RINA
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Prolapse; Female
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Posterior colporrhaphy: Medical records of women received concomitant posterior colporrhaphy for their pelvic organ prolapse repairs. Comparison will be made to compare preoperative and postoperative conditions.
  Interventions: Procedure: posterior colporrhaphy

INTERVENTIONS:
Procedure: posterior colporrhaphy — posterior colporrhaphy for rectocele.

SUMMARY:
Compare the changes of preoperative and postoperative posterior colporrhaphy.

DETAILED DESCRIPTION:
Introduction:

Concomitant posterior colporrhaphy was frequently used during pelvic organ prolapse repair.

Objectives:

To evaluate the correlation between the presence of bowel symptoms and s rectocele severity and elucidate the impact of posterior colporrhaphy on bowel functions.

Methods:

Medical records of all consecutive women who received concomitant posterior colporrhaphy for their pelvic organ prolapse repairs were reviewed. In general, all women were requested to answer bowel incontinence assessment questionnaires before and after surgery.

Possible results:

Differences in rectocele severities between the presence or absence of fecal incontinence, flatus incontinence, constipation, diarrhea or sensation of residual stool will be shown.

ELIGIBILITY:
Inclusion Criteria:

* women with pelvic organ prolapse planned to receive concomitant posterior colporrhaphy

Exclusion Criteria:

* Pregnancy

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with pelvic organ prolapse planned to receive concomitant posterior colporrhaphy
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with fecal incontinence | before the operation, postoperative one month and three months.
  Number of participants present the symptom
Number of participants with flatus | before the operation, postoperative one month and three months.
  Number of patients present the symptom
Number of participants with constipation | before the operation, postoperative one month and three months.
  Number of patients present the symptom
Number of participants with diarrhea | before the operation, postoperative one month and three months.
  Number of patients present the symptom
Number of participants with sensation of residual stool | before the operation, postoperative one month and three months.
  Number of patients present the symptom

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided